CLINICAL TRIAL: NCT01243606
Title: Efficacy Evaluation of a Unified Transdiagnostic Treatment for Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David H. Barlow, Professor of Psychology and Psychiatry, Emeritus. Founder and Director Emeritus, Center for Anxiety and Related Disorders at Boston University, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MH090053-01 (NIH)
Record Dates: First submitted 2010-11-12; First posted 2010-11-18 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Anxiety Disorders; Mood Disorders
Keywords: Anxiety; Depression; Obsessive Compulsive Disorder; Panic Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder; Transdiagnostic Treatment; CBT
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Depression; Obsessive-Compulsive Disorder; Panic Disorder; Generalized Anxiety Disorder; Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single Diagnosis Treatment Protocols (Experimental): Four disorder-specific cognitive-behavioral treatments will be conducted in accordance with treatment manuals of demonstrated efficacy. SDPs will be matched to the principal anxiety disorder diagnosis.
  Interventions: Behavioral: Single Diagnosis Treatment Protocol
- Unified Protocol (Experimental): The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders will be individually administered in accordance with a treatment protocol.
  Interventions: Behavioral: Unified Protocol (UP)
- Waitlist Control (No Intervention): Waitlist participants will not receive treatment during a 16-week waitlist period, but will receive the treatment of their choice immediately following the 16 week waiting period.

INTERVENTIONS:
Behavioral: Single Diagnosis Treatment Protocol — SDPs include: Managing Social Anxiety: A CBT Approach; Mastery of Anxiety and Panic-IV; Mastery of Anxiety and Worry-II; and Obsessive-Compulsive Disorder: A CBT Approach
  Arms: Single Diagnosis Treatment Protocols
Behavioral: Unified Protocol (UP) — The UP is designed to help patients learn how to confront and experience uncomfortable emotions and learn how to respond to their emotions in more adaptive ways. Individual treatment sessions will be conducted by experienced clinicians who will be trained in the administration of this protocol. A workbook will be provided to each patient as part of this manualized treatment. Treatment and session length of the UP will be matched to the SDPs for each principal diagnosis (see description above).
  Arms: Unified Protocol

SUMMARY:
Anxiety disorders are common, chronic, costly, debilitating to quality of life, and are more prevalent than any other class of disorders in every country in the world where surveys have been taken. Deepening understanding of the nature of anxiety and related emotional disorders during the last decade has revealed that commonalities in etiology and latent structure among these disorders supersedes differences. At the same time, examination of extant single diagnosis psychological treatment protocols (SDPs) for these disorders underscores mechanistic similarities. These findings suggested the possibility of distilling a set of psychological procedures that would comprise an innovative Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP), and this protocol has now been developed. If efficacious, the UP may represent a more efficient and possibly more effective strategy which would render treatment implications of comorbidity, not otherwise specified (NOS) and subdefinitional threshold anxiety disorder conditions moot.

The investigators now propose an evaluation of the efficacy of the UP in a group of patients with heterogeneous anxiety disorders by way of rigorous comparisons to existing evidence based SDPs benchmarked against a wait list control condition, using both statistical equivalence and superiority analyses. Additional aims include determining the durability of the UP relative to comparison conditions after treatment discontinuation, and ascertaining the differential impact of treatments on disorder specific symptoms vs. higher-order temperamental variables. Further analyses will indicate if changes in these higher order temperamental variables mediate long-term outcome as preliminary data suggests, and if this mechanism of action differs among treatments.

DETAILED DESCRIPTION:
The purpose of this proposal is to evaluate efficacy of the recently developed Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP). This protocol takes advantage of recent advances in our understanding of the nature of anxiety disorders, as well as emerging knowledge of the process of regulation and change in anxious behavior, in order to distill and refine basic principles of successful psychological treatments for anxiety disorders. It is expected that this approach will simplify training and dissemination, provide better coverage for comorbid conditions, cover "not otherwise specified" (NOS) and sub-definitional threshold presentations, possibly improve efficacy particularly in the long term, and perhaps also shed further light on the nature of anxiety disorders.

A heterogeneous sample of 250 patients meeting diagnostic criteria for at least one of four anxiety disorders: Social Phobia (SAD), Panic Disorder with or without Agoraphobia (PD/A), Generalized Anxiety Disorder (GAD), or Obsessive Compulsive Disorder (OCD) will be randomized to one of three treatment cells: (1) the Unified Protocol (UP); (2) a single diagnosis psychological treatment protocol (SDP); or (3) Wait List (WL). A minimum of 50 patients from each of the 4 principal diagnostic categories will be included in the randomization to ensure adequate representation of each anxiety disorder. The study will consist of two phases: (1) a 12 or 16 week acute treatment phase (or 16 week WL) and (2) a 12-month follow-up phase, during which active treatments will be discontinued and patients will be followed to assess the long-term effects of treatment (outcome measures are discussed below). Patients randomized to the WL condition will not enter the post-treatment period. Rather, they will be immediately assigned to their choice of either UP or SDP treatment at the end of the sixteen week waiting period.

All assessment and treatment procedures will be conducted at the Center for Anxiety and Related Disorders (CARD) at Boston University, which is one of the largest research clinics devoted to anxiety and related emotional disorders in the world. Total duration for participation in the study will not exceed 18 months total.

The major aims of this proposal are to:

Primary Aims

Aim 1: Evaluate the efficacy of the UP applied to a group of patients with heterogeneous anxiety disorders as compared to a group receiving existing evidence-based single diagnosis treatment protocols (SDPs) benchmarked against a wait list control condition (WL) to determine the treatment responsiveness of the sample on common measures of outcome.

Aim 2: Evaluate the efficacy of both the UP and SDPs relative to a benchmark WL condition.

Aim 3: Determine long-term efficacy of UP relative to SDPs over a 1-year period following treatment discontinuation.

Aim 4: Examine the relative effects of each active treatment approach (UP & SDPs) on comorbid anxiety and depressive disorder severity.

Secondary Aims

Aim 5: Ascertain the relative effects of each active treatment on higher-order temperamental indices.

Aim 6: Determine if change in higher order temperamental variables mediates long term outcome.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion, subjects will be males and females 18 years or older, fluent in the English language who have a principal DSM-IV diagnosis of SAD, PD/A, GAD, or OCD. In addition, to be eligible for participation, individuals must be willing to refrain from initiating additional treatment during the course of therapy unless mutually agreed upon with the therapists and the principal investigator; and willing to be randomly assigned to treatment conditions.

Exclusion Criteria:

* Patients will be excluded if they meet any of the following criteria:

  * Current DSM-IV diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, or organic mental disorder.
  * Clear and current suicidal risk.
  * Current or recent (past 90 days) history of substance abuse or drug dependence, with the exception of nicotine, marijuana, and caffeine.

Individuals will also be excluded if they previously received an adequate trial of CBT or if their emotional symptomatology is due to a medical/physical condition in which case alternative treatment would be clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule (ADIS): change over time | Baseline, every 4 weeks during a 16 week treatment or waitlist period, 6-month follow-up, 12-month follow-up
  The ADIS is a semi-structured diagnostic interview designed to establish reliable DSM anxiety, mood, somatoform and substance use disorders. For each current diagnosis, interviewers assigned a 0-8 clinical severity rating (CSR) that indicates their judgment of the degree of distress and impairment associated with the disorder (0=none to 8=very severely disturbing/disabling). The information derived from the interview using the ADIS allows clinicians to determine differential diagnoses and gain a clear understanding of the level and severity of each diagnosis.

SECONDARY OUTCOMES:
Clinical Global Impression Severity (CGI-S) and Improvement Scales (CGI-I): change over time | Baseline, Post-Treatment (approximately 16 weeks after Baseline) or Post-Wait List (16 weeks after Baseline), 6-month follow-up, 12-month follow-up
  These widely used clinician-rated instruments assess global severity and improvement from pre-treatment baseline on 7-point scales. The CGI-S and CGI-I will be used to define clinical response.
Structured Interview Guide for the Hamilton Anxiety and Depression Rating Scale (SIGH-A and SIGH-D): change over time | Baseline, Post-Treatment (approximately 16 weeks after Baseline) or Post-Wait List (16 weeks after Baseline),6-month follow-up, 12-month follow-up
  The SIGH-A and SIGH-D were developed to create a structured format for administering the Hamilton Anxiety Rating Scale (HARS; Hamilton, 1959) and the Hamilton Rating Scale for Depression (HRSD; Hamilton, 1960). Both include specific instructions on administration and anchor points for assigning severity ratings.
Yale-Brown Obsessive Compulsive Scale Interview-II (Y-BOCS-II): change over time | Baseline, Post-Treatment (approximately 16 weeks after Baseline) or Post-Wait List (16 weeks after Baseline),6-month follow-up, 12-month follow-up
Panic Disorder Severity Scale (PDSS): change over time | Baseline, Post-Treatment (approximately 16 weeks after Baseline) or Post-Wait List (16 weeks after Baseline),6-month follow-up, 12-month follow-up
Liebowitz Social Anxiety Scale (LSAS): change over time | Baseline, Post-Treatment (approximately 16 weeks after Baseline) or Post-Wait List (16 weeks after Baseline),6-month follow-up, 12-month follow-up
Generalized Anxiety Disorder Severity Scale (GADSS): change over time | Baseline, Post-Treatment (approximately 16 weeks after Baseline) or Post-Wait List (16 weeks after Baseline),6-month follow-up, 12-month follow-up
Overall Anxiety Sensitivity and Impairment Scale (OASIS)/ Overall Depression Sensitivity and Impairment Scale (ODSIS): change over time | Baseline, every 4 weeks during a 16 week treatment or waitlist period, Post-Treatment (12-16 weeks after Baseline) or Post-Wait List (16 weeks after Baseline), 6-month follow-up, 12-month follow-up
Work and Social Adjustment Scale (WSAS):change over time | Baseline, Post-Treatment (approximately 16 weeks after Baseline) or Post-Wait List (16 weeks after Baseline), 6-month follow-up, 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David H Barlow, Ph.D., Principal Investigator — Boston University
Locations (1):
- Center for Anxiety and Related Disorders at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cardona ND, Ametaj AA, Cassiello-Robbins C, Tirpak JW, Olesnycky O, Sauer-Zavala S, Farchione TJ, Barlow DH. Outcomes of People of Color in an Efficacy Trial of Cognitive-Behavioral Treatments for Anxiety, Depression, and Related Disorders: Preliminary Evidence. J Nerv Ment Dis. 2023 Sep 1;211(9):711-720. doi: 10.1097/NMD.0000000000001692. Epub 2023 Jul 10. PMID 37432031
- [Derived] Wilner Tirpak J, Cassiello-Robbins C, Ametaj A, Olesnycky OS, Sauer-Zavala S, Farchione TJ, Barlow DH. Changes in positive affect in cognitive-behavioral treatment of anxiety disorders. Gen Hosp Psychiatry. 2019 Nov-Dec;61:111-115. doi: 10.1016/j.genhosppsych.2019.06.008. Epub 2019 Jun 17. PMID 31253437
- [Derived] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327
- See also: Visit our website to learn more about the study. — http://bostonanxietytreatment.com